CLINICAL TRIAL: NCT04175691
Title: Clinical Significance of Circulating Non-coding RNA in Acute Ischemic Stroke (AISRNA)
Brief Title: Circulating Non-coding RNA in Acute Ischemic Stroke (AISRNA)
Acronym: AISRNA
Status: Recruiting | Type: Observational
Sponsor: Nanjing First Hospital, Nanjing Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: AISRNA
Record Dates: First submitted 2019-11-21; First posted 2019-11-25 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-11

CONDITIONS: Acute Stroke; Ischemic Stroke
Keywords: acute ischemic stroke; noncoding RNA; clinical significance; outcome
MeSH Terms: conditions — Stroke; Ischemic Stroke | interventions — Real-Time Polymerase Chain Reaction

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 90 Days
Biospecimen Retention: Samples With DNA — An 10 ml peripheral venous blood will be collected from the participants before and after interventions (i.e. intravenous thrombolysis and/or endovascular therapy)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- AIS group: This group includes patients with acute ischemic stroke (AIS).
  Interventions: Genetic: Sequencing of circRNA/miRNA/lncRNA
- HC group: This group includes healthy controls (HC).
  Interventions: Genetic: Sequencing of circRNA/miRNA/lncRNA

INTERVENTIONS:
Genetic: Sequencing of circRNA/miRNA/lncRNA — Next generation sequencing of circular RNA (circRNA), micro-RNA (miRNA) and long non-coding RNA (lncRNA)
  Other Names: Quantitative Real-time polymerase chain reaction

SUMMARY:
AISRNA is to analyze the expression pattern of circular RNA (circRNA), micro-RNA (miRNA) and long non-coding RNA (lncRNA) by next-generation sequencing in patients with acute ischemic stroke and healthy control. The candidate circRNA/miRNA/lncRNA will be verified as biomarkers for the detection and prognosis of acute ischemic stroke.

DETAILED DESCRIPTION:
Noncoding RNAs have been highlighted to be involved in the pathological process of ischemic stroke (IS). The purpose of this protocol will investigate the expression pattern of circular RNA (circRNA), micro-RNA (miRNA) and long non-coding RNA (lncRNA) by next-generation sequencing in patients with acute ischemic stroke and healthy control. The candidate circRNA/miRNA/lncRNA will be verified as biomarkers for the detection and prognosis of acute ischemic stroke. Distinctive expression patterns of circRNA/miRNA/lncRNA will be identified by the next-generation sequencing and individual quantitative real time polymerase chain reaction (qRT-PCR). A diagnostic or predictive model will be established using logistic regression. The panel of these altered ncRNAs may be associated with acute IS and could serve as a novel diagnostic or predictive method.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or older
* Confirmed acute ischemic stroke by a diffusion-weighted imaging-position lesion on magnetic resonance imaging (MRI) and a new lesion on a brain computed tomography (CT) scan
* Within 72 hours of symptom onset
* Good performance status
* Signed an approved informed consents

Exclusion Criteria:

-a history of hemorrhagic infarction, chronic kidney/liver diseases, peripheral arterial occlusive disease, active malignant disease, and inflammatory or infectious diseases

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: There will be 5 AIS patients and 5 HCs, whose data will be applied for construction of diagnostic and predictive models of circRNA/miRNA/lncRNA from the circulating blood. There will be 100 patients suspected of AIS (such as transient ischemic attack) 300 AIS patients, whose data will be applied for validation of such diagnosis and predictive models, respectively.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2019-11-24 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Differential expression pattern of circRNA/miRNA/lncRNA | 90 days
  Differential expression pattern of circular RNA (circRNA), micro-RNA (miRNA) and long non-coding RNA (lncRNA) will be compared between AIS group and HC group, thus candidate circRNA/miRNA/lncRNA will be verified as biomarkers for the detection and prognosis of AIS.

SECONDARY OUTCOMES:
Prognostic value of circRNA/miRNA/lncRNA in acute ischemic stroke | 90 days
  The prognosis of AIS patients will be analyzed between differential expressed candidate miRNA/lncRNA after they have completed the systematic therapy.
Correlation of circRNA/miRNA/lncRNA and inflammatory factors in acute ischemic stroke | 7 days
  Correlation of circRNA/miRNA/lncRNA and inflammatory factors on admission will be explored in acute ischemic stroke.
Correlation of circRNA/miRNA/lncRNA and stroke-associated infection | 30 days
  Correlation of circRNA/miRNA/lncRNA and stroke-associated infection will be explored in acute ischemic stroke.
Dynamic changes of circRNA/miRNA/lncRNA during the follow-up period | 90 days
  Dynamic changes of circRNA/miRNA/lncRNA will be explored before and after endovascular therapy

CONTACTS AND LOCATIONS:
Overall Officials: Junshan Zhou, Professor, Study Chair — Nanjing Medical University
Locations (1):
- Nanjing First Hospital, Nanjing Medical University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Yes
All information will be available to all researchers.
Supporting Information: Study Protocol
Time Frame: All information will be available to all researchers when related investigation has been accepted publicly, and will be available for 5 years.
Access Criteria: All information will be available to all researchers when related investigation has been accepted publicly.

REFERENCES:
- [Background] Deng QW, Li S, Wang H, Sun HL, Zuo L, Gu ZT, Lu G, Sun CZ, Zhang HQ, Yan FL. Differential long noncoding RNA expressions in peripheral blood mononuclear cells for detection of acute ischemic stroke. Clin Sci (Lond). 2018 Jul 31;132(14):1597-1614. doi: 10.1042/CS20180411. Print 2018 Jul 31. PMID 29997237
- [Background] Li S, Lu G, Wang D, He JL, Zuo L, Wang H, Gu ZT, Zhou JS, Yan FL, Deng QW. MicroRNA-4443 regulates monocyte activation by targeting tumor necrosis factor receptor associated factor 4 in stroke-induced immunosuppression. Eur J Neurol. 2020 Aug;27(8):1625-1637. doi: 10.1111/ene.14282. Epub 2020 May 18. PMID 32337817
- [Derived] Chen W, Zhang H, Li Z, Deng Q, Wang M, Chen Y, Zhang Y. Effects of edaravone dexborneol on functional outcome and inflammatory response in patients with acute ischemic stroke. BMC Neurol. 2024 Jun 20;24(1):209. doi: 10.1186/s12883-024-03712-1. PMID 38902691
- [Derived] Sun H, Li S, Xu Z, Liu C, Gong P, Deng Q, Yan F. SNHG15 is a negative regulator of inflammation by mediating TRAF2 ubiquitination in stroke-induced immunosuppression. J Neuroinflammation. 2022 Jan 3;19(1):1. doi: 10.1186/s12974-021-02372-z. PMID 34980176
- [Derived] Deng QW, Huang S, Li S, Zhai Q, Zhang Q, Wang ZJ, Chen WX, Sun H, Lu M, Zhou J. Inflammatory Factors as Potential Markers of Early Neurological Deterioration in Acute Ischemic Stroke Patients Receiving Endovascular Therapy - The AISRNA Study. J Inflamm Res. 2021 Sep 2;14:4399-4407. doi: 10.2147/JIR.S317147. eCollection 2021. PMID 34511974
- See also: Differential Long Noncoding RNA Expressions in Peripheral Blood Mononuclear Cells for Detection of Acute Ischemic Stroke — http://pubmed.ncbi.nlm.nih.gov/29997237/